CLINICAL TRIAL: NCT05959655
Title: Modern Urodynamics System Efficacy (MUSE) Study
Acronym: MUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bright Uro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-0005
Record Dates: First submitted 2023-07-07; First posted 2023-07-25 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Urologic Diseases; Urodynamics
Keywords: Lower Urinary Tract Dysfunction; Urinary Incontinence; Overactive Bladder; Urodynamics; Uroflowmetry
MeSH Terms: conditions — Urologic Diseases; Urinary Incontinence; Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Glean Urodynamics System (Experimental): Wireless, catheter-free urodynamics system
  Interventions: Device: Glean Urodynamics System

INTERVENTIONS:
Device: Glean Urodynamics System — Wireless, catheter-free urodynamics system
  Other Names: GUS

SUMMARY:
The goal of this prospective trial is to evaluate the feasibility, efficacy, and safety of the Glean Urodynamics System (GUS) for use in the clinic to collect vesical pressure data in adult males and females with lower urinary tract symptoms.

The main question[s] it aims to answer are:

• What is the feasibility, efficacy, and safety of GUS for use in clinical to collect vesical pressure data in adult males and females with lower urinary tract symptoms?

Participants will undergo a planned conventional urodynamics exam after which the Glean Sensor will be inserted and ambulatory urodynamics will be performed with the sensor indwelling in the bladder after which the sensor will be removed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient must be ≥ 18 years of age
* Patient must have a diagnosis of LUTD
* Patient must be scheduled for or recommended for cUDS
* Patient is able to tolerate 18Fr catheterization
* Patient or patient's legally authorized representative is able to provide informed consent

Exclusion Criteria:

* Pregnant (as confirmed by urine pregnancy test) or breastfeeding, pregnant within the past 6 months or intend to become pregnant during the study period.
* Patient has a symptomatic UTI based on CDC guidance (see below)
* Subjects who, at the principal investigator's determination, would not be appropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Carter, DHSc, MPH, Study Director — Bright Uro
Locations (5):
- United States (5):
  - Tri Valley Urology, Murrieta, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stony Brook Medicine, East Setauket, New York
  - Palmetto Adult and Children's Urology, North Charleston, South Carolina
  - Urology Partners of North Texas, Arlington, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frainey BT, Majerus SJA, Derisavifard S, Lewis KC, Williams AR, Balog BM, Butler RS, Goldman HB, Damaser MS. First in Human Subjects Testing of the UroMonitor: A Catheter-free Wireless Ambulatory Bladder Pressure Monitor. J Urol. 2023 Jul;210(1):186-195. doi: 10.1097/JU.0000000000003451. Epub 2023 Jun 9. PMID 37293725
- [Result] Kim J, Xavier K, Cannon-Smith T, Vaughan T, Vemulapalli S, Zhao H, Aalami-Harandi A, Shah N. The Feasibility and Safety of the Glean Urodynamics System: The Modern Urodynamics System Efficacy Study. J Endourol. 2025 Jun;39(6):625-634. doi: 10.1089/end.2025.0270. Epub 2025 May 2. PMID 40314068

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glean Urodynamics System
Started | 38
Underwent Conventional UDS | 34
Underwent Glean Urodynamics | 32
Completed | 28
Not Completed | 10

BASELINE CHARACTERISTICS:
Population: Participants enrolled in the study
Arm/Group | Glean Urodynamics System
Number analyzed (Participants) | 38
Age, Customized [Mean (Full Range); unit: Years]
  Age | 64 [25 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Insertion Success
Description: Percent of insertion attempts of the Glean sensor deemed successful
Time Frame: during the insertion procedure of a device
Population: 33/34 participants who underwent conventional urodynamics underwent an insertion attempt with the Glean Urodynamics System.
Measure: Count of Participants; unit: Participants
Arm/Group | Glean Urodynamics System
Number analyzed (Participants) | 33
Participants | 32

2. Primary Outcome: Percentage of Participants With a Device-related SAE
Description: Device-related serious adverse events
Time Frame: up to 2 weeks
Population: Number of participants undergoing Glean Urodynamics
Measure: Count of Participants; unit: Participants
Arm/Group | Glean Urodynamics System
Number analyzed (Participants) | 32
Participants | 0

3. Secondary Outcome: Percentage of Participants Rating Overall Comfort of Glean Urodynamics as Comfortable or Extremely Comfortable
Description: Number of participants rating the overall comfort of Glean Urodynamics at comfortable or extremely comfortable
Time Frame: asked at end of Glean Urodynamics procedure
Population: Number of participants who experienced Glean Urodynamics and completed the survey at the end of the urodynamics study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Glean Urodynamics System
Number analyzed (Participants) | 31
Participants | 13

4. Primary Outcome: Percentage of Participants With Removal Success
Description: Percent of removal attempts of the Glean sensor deemed successful
Time Frame: during the removal procedure of a device
Population: 32 participants had Glean successfully inserted and thus all had a successful removal.
Measure: Count of Participants; unit: Participants
Arm/Group | Glean Urodynamics System
Number analyzed (Participants) | 32
Participants | 32

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 2 weeks
Groups:
- All Participants: All participants enrolled in the study
- Glean Urodynamics System: Among those who underwent Glean Urodynamics
Arm/Group | All Participants | Glean Urodynamics System
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/32
Other Adverse Events (participants affected / at risk) | 12/38 | 7/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=38) | Glean Urodynamics System (N=32)
Gross Hematuria (Renal and urinary disorders) | 9 (9) | 4 (4)
Genitourinary pain or discomfort (Renal and urinary disorders) | 2 (2) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Study not powered for any outcome or any comparisons; small sample size limits validity, generalizability, and applicability; order of procedures (i.e., conventional UDS occurring before Glean UDS) and the variability of standard-of-care may have influenced results such as attribution of harm; and participant recall bias due to the removal of the Glean sensor being the last procedure experienced (Kim, 2025).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT05959655/Prot_SAP_000.pdf